CLINICAL TRIAL: NCT05431985
Title: Cross-cultural Validation of a Screening Scale for the Misuse of Opioid Analgesics in Primary Care
Acronym: VAMOS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2015 LAPORTE
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Chronic Pain; Addiction Opiate
Keywords: chronic pain; opioids; primary care; misuse; addiction
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: Analgesic Opioids misuse among patients with chronic pain ranges from 0% to 50%. The general practitioner is the first prescriber of opioid analgesics Our objective was to validate in primary care the POMI (Prescription Opioid Misuse Index) to identify the misuse of AOs.

Study Setting: Patients with chronic pain, taking AOs for at least 3 months, and followed in general practice.

Study design: Psychometric study

Data Collection/Extraction methods: Eligible patients followed in general practice responded to the POMI: Test phase. They then responded after 2 weeks: the retest. The gold standard used was the DSM-V.

DETAILED DESCRIPTION:
Chronic pain represents a major problem in terms of individual, quality of life, and collective impact: cost generated by delays in treatment and care. The prevalence of chronic pain among the general population varies from 10.1 to 55.2%. In the front line, general practitioners (GP) are at the heart of treating pain : pain represent 43% of the reasons for the consultation, 24% of these being for chronic pain. More than half of these patients had exclusive care through their GP. The others are followed up in a pain assessment and treatment center.

In 2015, nearly one in five French people (17,1%) of French people have taken opioid treatment. The risk of opioid use disorder secondary to opioid analgesics among patients suffering from chronic pain varies from 0% to 50%. American recommendations advocate periodic surveillance of this opioid use disorder depending on the patient's risk factors, when chronic opioid analgesics are prescribed. The French "Limoges" recommendations also mention a systematic search for signs of psychological dependence during treatment and state that treatment with strong opioids should be stopped in the event of misuse, abuse or addiction. They recommend, on each examination, the investigation for signs of misuse or psychological dependence (characterised by craving) as ways of monitoring that strong opioids are being correctly used in chronic osteo-articular pain.

Identifying the misuse is a way of optimising their benefit/risk ratio

The difficulty in establishing the prevalence of misuse is due to a lack of standardization of studies and the lack of consensus in the use of assessment tools. Several tools are available internationally. The only diagnostic criteria available are those of the DSM-5 (Fifth Edition of the Diagnostic and Statistical Manual of Mental Disorders) or the ICD-10 which overestimate this prevalence notably by the presence of frequent tolerance and withdrawal criteria for these patients, in the absence of misuse or addiction. Today, no screening scale has been validated in France for primary care, but recently, the authors have validated the POMI scale in French to screen the patients specifically followed in pain clinic and presenting a misuse behavior of their opioid analgesic treatment. In 2015, treatment initiation was carried out by a GP in 59.1% of cases for weak opioid and 62.9% of cases for strong opioids and by a hospital doctor for 20.1% and 21% respectively7. Currently, no scale was validated in primary care. A scale validated in French would make it possible to standardize these screening practices and secure prescription both from the point of view of the doctor and of the patient. Furthermore, this absence of a validated tool in French is proving to be an obstacle to the development of true pharmaco-epidemiological studies on the prevalence of the opioids misuse. The originality of this study is to assess the clinical relevance of the french transcultural validation of the POMI scale in primary care in order to ensure an appropriate and relevant use by all health professionals and to allow large-scale screening for the misuse behavior of analgesic opioids.

The aim of the study was a validation of the French version of the Prescription Opioid Misuse Index - POMI patients with chronic pain in general practitioners setting.

Secondary objective

* To study the profile of participants with misuse of opioid analgesics.
* To compare the results of this study with the previous study on patients followed in pain clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over,
* Patients with chronic pain for at least 6 months,
* Patients with a prescription from the GP of at least one Opioid analgesic drug taken daily for at least the previous 3 months,
* Patients registered with the French insurance system.

Exclusion Criteria:

* Discontinuation of opioid prescriptions on the test phase day (no Retest possible),
* Patients in the process of withdrawal (risk of having been withdrawn during the Retest phase),
* Patients unable to complete the questionnaire alone,
* Patients who are monitored by a pain clinic or addiction centre,
* Patients with ongoing cancer,
* Patients refusing to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with chronic pain for at least 6 months, and with a prescription from the general practitioners of at least one opioid analgesic drug taken daily for at least the previous 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Prescription Opioid Misuse Index - POMI | at inclusion
  Prescription Opioid Misuse Index (POMI) scale was developed in the United States to assess the oxycodone misuse. This scale was validated among 137 subjects recruited from pain clinics, addiction treatment programs, jails, or private medical practice. The POMI is an 8 point self-assessment scale each numbered 0 (absence) or 1 (presence). The sum of point is used to calculate a score (between 0 and 8) and a score of more or equal to 2 is considered as positive and describe a misuse.
Prescription Opioid Misuse Index - POMI | 2 weeks after the first completion
  Prescription Opioid Misuse Index (POMI) scale was developed in the United States to assess the oxycodone misuse. This scale was validated among 137 subjects recruited from pain clinics, addiction treatment programs, jails, or private medical practice. The POMI is an 8 point self-assessment scale each numbered 0 (absence) or 1 (presence). The sum of point is used to calculate a score (between 0 and 8) and a score of more or equal to 2 is considered as positive and describe a misuse.

SECONDARY OUTCOMES:
Sociodemographic characteristics | once, at inclusion
  GPs asked patients about sociodemographic data (age, gender, family status, professional status); medical and family medical history; history of psychiatric problem, substance use and abuse.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Clermont-Ferrand, UMR INSERM 1107, NEURO-DOL, Clermont-Ferrand
  - Département de médecine Générale, Facultés de Médecine de Clermont-Ferrand, Clermont-Ferrand
  - Département de médecine générale, Lyon, Lyon
  - Département de médecine générale, Faculté de médecine, Montpellier, Montpellier
  - Département de médecine générale, Faculté de médecine, Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No